CLINICAL TRIAL: NCT04652908
Title: Phase 1/2a Trial of Placental Mesenchymal Stem Cells for Repair of Fetal Myelomeningocele
Brief Title: Cellular Therapy for In Utero Repair of Myelomeningocele - The CuRe Trial
Acronym: CuRe
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1617774
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Myelomeningocele
MeSH Terms: conditions — Meningomyelocele

STUDY DESIGN:
Intervention Model Description: Treatment arm subjects receiving PMSC-ECM (Placental Mesenchymal Stem Cells seeded on a commercially available dural graft extracellular matrix). Additionally, we will follow a contemporaneous cohort of patients undergoing routine fetal or postnatal MMC repair without PMSC-ECM (non-PMSC untreated contemporaneous cohort). 35 participants will be enrolled under the treatment arm and 20 participants will be enrolled under the untreated contemporaneous cohort.
  The addition of a non-PMSC treated cohort, the untreated contemporaneous cohort, has been added at the request of the FDA to provide contemporaneous patients for validation of the continued relevance of use of the outcomes of the MOMS trial as the comparison arm for the Phase 2a portion of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment with PMSC-ECM (Experimental): One-time administration of PMSC-ECM during the course of in utero fetal myelomeningocele surgery will be administered
  Interventions: Biological: Placental Mesenchymal Stem Cells seeded on a commercially available dural graft extracellular matrix
- non-PMSC untreated contemporaneous cohort (Other): Contemporaneous cohort of patients undergoing routine fetal or postnatal MMC repair without PMSC-ECM (non-PMSC untreated contemporaneous cohort).
  Interventions: Other: Untreated contemporaneous cohort

INTERVENTIONS:
Biological: Placental Mesenchymal Stem Cells seeded on a commercially available dural graft extracellular matrix — As in the current standard fetal surgery, under sonographic guidance, initial uterine entry will be accomplished by uterine stapling device or similar. The fetus will be given an intramuscular injection of pain medications and paralytic. The myelomeningocele will be closed in a standardized manner under magnification. As in the standard fetal operation, the spinal cord will be dissected from surrounding tissue and allowed to drop into the spinal canal. The PMSC-ECM product will then be tailored to the size of the spinal cord and applied topically, cell side down. The PMSC-ECM product will be sutured in place to the dura. Finally, the fetal skin will be closed in the standard fashion. The amniotic fluid volume will be replaced and antibiotics will be added. The uterus will be closed. The abdominal fascial layer and skin will be closed in routine fashion.
  Other Names: PMSC-ECM
  Arms: Treatment with PMSC-ECM
Other: Untreated contemporaneous cohort — The addition of a non-PMSC treated cohort, the untreated contemporaneous cohort, has been added at the request of the FDA to provide contemporaneous patients for validation of the continued relevance of use of the outcomes of the MOMS trial as the comparison arm for the Phase 2a portion of the study.
  Other Names: non-PMSC-ECM
  Arms: non-PMSC untreated contemporaneous cohort

SUMMARY:
Spina bifida, or myelomeningocele (MMC), is a birth defect that results in paralysis, excess fluid on the brain (hydrocephalus), and impaired ability to urinate and have bowel movements normally. In a previous study (the MOMS trial), surgery before birth (in-utero/fetal surgery) was shown to reduce the need for shunting for hydrocephalus. There was also some improvement in ambulation, but 58 % of the children still could not walk unassisted.

This study is testing living stem cells from placenta added to the fetal repair in an effort to improve the ability to walk. Previous animal studies have shown dramatic improvement in walking and bowel and bladder function when placental stem cells are added to MMC repair. Use of these "living" cells may protect the developing spinal cord, prevent further injury, and may even reverse existing damage to the nerves that control movement. This study is assessing the safety and efficacy of adding stem cells to open fetal surgery for MMC in humans.

DETAILED DESCRIPTION:
Historically, treatment of MMC was limited to post-natal surgery to close the dura and skin over the spinal cord to prevent meningitis, which had no effect on motor function. The potential benefit of earlier intervention was realized when prenatal ultrasound of patients with MMC early in gestation revealed near-normal leg movements despite displaying paralysis at birth. This finding gave credence to the two-hit hypothesis that paralysis was progressive during prenatal life and suggested that fetal intervention could prevent the secondary damage to the spinal cord. Fetal repair of MMC did confer improvement in motor function of children treated in the Management of Myelomeningocele (MOMS) randomized controlled trial. The promising results of the MOMS trial demonstrated the potential for improvement of paralysis for these patients, but distal motor function still remained severely impaired in the majority of patients with MMC with standard in utero repair alone. While this demonstrated that the ideal time to intervene to prevent paralysis is in utero with the goal of preventing the accrual of ongoing damage to the spinal cord, there is still room for improvement. The remarkable regenerative capacity of the fetal environment combined with regenerative capacity of placental mesenchymal stem cells offers potential for augmentation of the fetal repair of MMC with a novel therapy to further reduce and repair the sustained spinal cord damage.

ELIGIBILITY:
Inclusion Criteria:

Eligibility for fetal surgery per the MOMS trial, which are:

* Myelomeningocele (including myeloschisis) at any level from T1 through S1 with hindbrain herniation. Lesion level will be confirmed by ultrasound and hindbrain herniation will be confirmed by MRI at the UC Davis Fetal Center
* Maternal age ≥18 years
* Gestational age at enrollment between 19 weeks 0 days and 25 weeks 6 days gestation as determined by clinical information and evaluation of first ultrasound
* Normal karyotype. Results by fluorescence in situ hybridization (FISH) will be acceptable if the patient is greater than 24 weeks gestation;

Exclusion Criteria:

Not being eligible for fetal surgery per the MOMS trial, which includes:

* Multifetal pregnancy
* Insulin dependent pregestational diabetes
* Fetal anomaly not related to myelomeningocele.
* Kyphosis in the fetus of 30 degrees or more
* Current or planned cerclage or documented history of incompetent cervix, placenta previa or placental abruption
* Short cervix < 20 mm measured by cervical ultrasound
* Obesity as defined by body mass index of 35 or greater
* Previous spontaneous singleton delivery prior to 37 weeks
* Maternal-fetal Rh isoimmunization, Kell sensitization or a history of neonatal alloimmune thrombocytopenia
* Maternal HIV or Hepatitis-B status positive due to the increased risk of transmission to the fetus during maternal-fetal surgery. If the patient's HIV or Hepatitis B status is unknown, the patient must be tested and found to have negative results before she can be enrolled
* Known Hepatitis-C positivity. If the patient's Hepatitis C status is unknown, she does not need to be screened
* Uterine anomaly such as large or multiple fibroids or Müllerian duct abnormality
* Other maternal medical condition which is a contraindication to surgery or general anesthesia. This includes any patient with a previous hysterotomy in the active segment of the uterus (whether from a previous classical cesarean, uterine anomaly such as an arcuate or bicornuate uterus, major myomectomy resection, or previous fetal surgery)
* Patient does not have a support person (e.g., husband, partner, mother)
* Inability to comply with the travel and follow-up requirements of fetal surgery
* Patient does not meet other psychosocial criteria (as determined by the psychosocial interviewer) to handle the implications of fetal surgery
* Participation in another intervention study that influences maternal and fetal morbidity and mortality or participation in this trial in a previous pregnancy;
* Maternal hypertension which would increase the risk of preeclampsia or preterm delivery (including, but not limited to: uncontrolled hypertension, chronic hypertension with end organ damage and new onset hypertension in current pregnancy)
* Active COVID-19 infection at time of fetal surgery as determined by positive test

Ages: 19 Weeks to 25 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Estimated)
Dates: Start 2021-06-21 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Safety of the placenta-derived mesenchymal stem cell (PMSC-ECM) Product | Assessed at birth
  Will be assessed by evaluating the presence or absence of cerebrospinal fluid leak, infection at the MMC repair site, failure of the MMC repair site to heal, and any unexpected growths or tumor formation. These will be assessed at birth by physical exam, brain and spinal ultrasound , and brain and spinal MRI.

SECONDARY OUTCOMES:
Efficacy of the PMSC-ECM Product | 30 months.
  This is primarily evaluated by improvement in motor function 2 or more levels greater than expected by anatomic level of the defect and by patients' ability to walk independently. Bowel function will be assessed by caregiver questionnaires on bowel habits, and by anorectal manometry. Urologic function will be assessed by caregiver questionnaires regarding urologic function, by renal and bladder ultrasounds to evaluate for hydronephrosis and bladder abnormalities, and by video urodynamics.

CONTACTS AND LOCATIONS:
Overall Officials: Diana L Farmer, MD, Principal Investigator — UC Davis School of Medicine
Locations (1):
- UC Davis Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No